CLINICAL TRIAL: NCT05562622
Title: Clinical Assessment of DOT Spectacle Lenses in Chinese Children
Brief Title: Assessment of DOT Spectacles in Chinese Children
Acronym: CATHAY
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: SightGlass Vision, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CPRO-2201-001
Record Dates: First submitted 2022-09-28; First posted 2022-10-03 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Juvenile Myopia; Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Evaluator/Investigational site staff tasked with measuring key primary variables (i.e., axial length and SER) will be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- SightGlass Vision Test Arm 1 (Experimental): Single vision, impact-resistant spectacle lenses
  Interventions: Device: Novel spectacle lens design
- Test Arm 2 (Other): Single vision, impact-resistant spectacle lenses
  Interventions: Device: Spectacle lenses

INTERVENTIONS:
Device: Novel spectacle lens design — Use of lenses may reduce the rate of progression of juvenile myopia
  Arms: SightGlass Vision Test Arm 1
Device: Spectacle lenses — Use of lenses may reduce the rate of progression of juvenile myopia
  Arms: Test Arm 2

SUMMARY:
This is a randomized, controlled, evaluator-blinded, multicenter, two-arm parallel group clinical trial of 12-months duration to evaluate the continued safety and efficacy of Diffusion Optics Technology (DOT) spectacle lenses by comparing to single vision, impact-resistant spectacle lenses in reducing the progression of juvenile myopia in children of Chinese origin.

ELIGIBILITY:
Inclusion Criteria:

1. Children 6-13 years of age
2. SER error between -0.75D and -5.00D
3. Willingness to wear study spectacles and participate in the trial for 12 months without contact lens wear

Exclusion Criteria:

1. Prior usage of atropine, multifocal contact lenses, or orthokeratology (ortho-K)
2. Astigmatism worse than -1.50 DC (by manifest refraction) in either eye
3. Anisometropia (SER manifest refraction) greater than 1.00 D

Ages: 6 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 195 (Actual)
Dates: Start 2023-02-05 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Axial length | 12 months
  Change in axial length from baseline

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - Aier Eye Hospital, Changsha
  - West China Hospital, Chengdu
  - Zhongshan Ophthalmic Center, Guangzhou
  - Fudan University EENT, Shanghai
  - Tianjin Eye Hospital, Tianjin